CLINICAL TRIAL: NCT01188447
Title: Evaluation of the Safety of C-Spine Clearance by Paramedics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009142-01H
Record Dates: First submitted 2010-08-20; First posted 2010-08-25 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Fracture of Cervical Spine
Keywords: cervical-spine injuries; cervical-spine fractures; spinal cord injury; neck injury; Canadian C-Spine Rule; paramedics; emergency medical services
MeSH Terms: conditions — Spinal Cord Injuries; Neck Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eligible low-risk trauma patients (Experimental): Paramedics will use the Canadian C-Spine Rule to evaluate low-risk trauma patients meeting the study inclusion criteria in order to determine the need for spinal immobilization for transport to the hospital.
  Interventions: Procedure: Canadian C-Spine Rule

INTERVENTIONS:
Procedure: Canadian C-Spine Rule — Paramedics will apply a validated decision rule (the Canadian C-spine Rule) to determine whether or not immobilization is required for trauma patients being transported to the emergency department.

SUMMARY:
The goal of this cohort study is to evaluate the safety and potential impact of an active strategy that allows paramedics to assess very low-risk trauma patients with the Canadian C-Spine Rule (CCR) and transport them to the Emergency Department without immobilization. The specific objectives of the study are to determine safety, determine the clinical impact and evaluate performance.

ELIGIBILITY:
Inclusion Criteria:

* consecutive alert, stable adults evaluated by the paramedics with potential c-spine injury after sustaining acute blunt trauma. Patient eligibility will be determined at the time of paramedic arrival at the scene based on the following criteria:
* "Potential c-spine injury after sustaining acute blunt trauma" will include patients with either:

  * neck pain with any mechanism of injury (subjective complaint by the patient of any pain in the posterior aspect of the neck),
  * no neck pain but some visible injury above the clavicles, and/or
  * neither neck pain nor visible injury, but significant mechanism of injury as determined by the paramedic at the scene.
* "Alert" is defined as a Glasgow Coma Scale score of 15 (converses, fully oriented, and follows commands).
* "Stable" refers to normal vital signs(systolic blood pressure 90 mm Hg or greater and respiratory rate between 10 and 24 breaths per minute).
* "Acute" refers to injury within the past 4 hours.

Exclusion Criteria:

* Patients under the age of 16 years,
* Patients with penetrating trauma from stabbing or gunshot wound,
* Patients with acute paralysis (paraplegia, quadriplegia),
* Patients with known vertebral disease (ankylosing spondylitis, rheumatoid arthritis, spinal stenosis, or previous cervical spine surgery), or
* Patients referred from another hospital and transported between facilities.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4034 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Paramedic Service, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaillancourt C, Charette M, Kasaboski A, Maloney J, Wells GA, Stiell IG. Evaluation of the safety of C-spine clearance by paramedics: design and methodology. BMC Emerg Med. 2011 Feb 1;11:1. doi: 10.1186/1471-227X-11-1. PMID 21284880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eligible Low-risk Trauma Patients
Started | 4034
Completed | 4034
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eligible Low-risk Trauma Patients
Number analyzed (Participants) | 4034
Age, Continuous [Mean (Full Range); unit: years] | 43 [16 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2150
  Male | 1884
Region of Enrollment [Number; unit: participants]
  Canada | 4034

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Measures of safety will include:
  1. number of missed cervical spine injuries
  2. number of serious adverse outcomes
Time Frame: within 30 days of enrollment
Measure: Number; unit: Adverse event
Arm/Group | Eligible Low-risk Trauma Patients
Number analyzed (Participants) | 4034
Adverse event | 1

2. Secondary Outcome: Clearance Rate
Description: Proportion of eligible low-risk patients transported without immobilization
Time Frame: Measures of clinical impact will be assessed immediately following the patient's Emergency Department visit
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: eligible patients evaluated with the Canadian C-Spine Rule
Arm/Group | Eligible Patients
Number analyzed (Participants) | 4034
Participants | 2569

3. Secondary Outcome: Performance of the Canadian C-Spine Rule
Description: Measurements of the performance of the rule will include:
  1. rule accuracy
  2. paramedic accuracy of interpretation
  3. paramedic agreement and level of comfort with the decision suggested by the Canadian C-Spine Rule
Time Frame: Rule accuracy will be within 30 days of enrollment. Paramedic accuracy of interpretation and agreement will be assessed immediately following enrollment.
Measure: Number (95% Confidence Interval); unit: percentage of injuries identified
Arm/Group | Eligible Low-risk Trauma Patients
Number analyzed (Participants) | 4034
percentage of injuries identified | 91 [58 to 100]

4. Secondary Outcome: Scene Time
Description: Time spent at scene (difference between Paramedic scene departure and arrival at patient side)
Time Frame: immediately following evaluation
Population: In order to be included in this analysis, a valid time for paramedic arrival and paramedic scene departure were required. Any patient refusing transport or missing time information was not included in the analysis.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Eligible Low-risk Trauma Patients
Number analyzed (Participants) | 3,174
Minutes | 18 [1 to 147]

5. Secondary Outcome: Average Contact Time
Description: Total time spent with patient (Defined as difference between Transfer of Care and Arrival at Patient Side)
Time Frame: immediately following evaluation
Population: In order to be included in this analysis, and to have Contact Time calculated, both the paramedic arrival time and transfer of care time were required. Any case missing this information could not be included in the calculation.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Eligible Low-risk Trauma Patients
Number analyzed (Participants) | 3,175
minutes | 55 [5 to 428]

ADVERSE EVENTS:
Arm/Group | Eligible Low-risk Trauma Patients
Serious Adverse Events (participants affected / at risk) | 0/4034
Other Adverse Events (participants affected / at risk) | 1/4034
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eligible Low-risk Trauma Patients (N=4034)
Missed C-Spine Injury (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No